CLINICAL TRIAL: NCT05496023
Title: Pre-stenting Angiography-derived Fractional Flow Reserve Pullback Guided PercutaneouS Coronary Intervention Predicts Physiological and Clinical Outcomes in Coronary Artery Disease
Brief Title: Angiography-derived FFR GPS in Predicting Post-PCI Physiological and Clinical Outcomes
Acronym: Angio-GPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS20220808; CHART2022-04 (Registry Identifier: CHART Angio-FFR GPS)
Record Dates: First submitted 2022-08-07; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre PCI state: The current study will analyze the angio-FFR and generate the virtual pullback. The pullback will be co-registered by overlaying the pullback onto coronary angiogram.
  Interventions: Device: Percutaneous coronary intervention
- Post-PCI state: The post-PCI FFR and angio-FFR will be meaured.

INTERVENTIONS:
Device: Percutaneous coronary intervention — 1. Pre-PCI angio-FFR was calculated and virtual pullback was generated
  2. Automated algorithm to calculate delta angio-FFR per unit length and co-registered onto coronary angiogram was developed
  3. PCI was performed using 2nd generation DES
  Groups: Pre PCI state

SUMMARY:
To investigate the feasibility of physiological map generated from angiography-derived fractional flow reserve (FFR) (angio-FFR) pullback and its value in predicting physiological and clinical outcomes after stenting.

DETAILED DESCRIPTION:
Physiological coronary lesion evaluation such as fractional flow reserve (FFR) is now recommended by guidelines to guide percutaneous coronary intervention (PCI). However, it was not widely used in subsequent years for a variety of reasons, including the additional time needed to measure pressure wire-derived FFR, technical challenges and the small risk associated with maneuvering a pressure wire down a coronary artery, the added time to assess multiple vessels, issues with drift in the pressure wire reading, and the time, expense, and associated side effects with some hyperemic agents necessary to measure FFR.

In recent years, advancements in technology made it possible to calculate FFR from conventional coronary angiography without the need of a pressure wire or hyperemic agent. The FAVOR III (Comparison of Quantitative Flow Ratio Guided and Angiography Guided Percutaneous InterVention in Patients With cORonary Artery Disease) China has demonstrated that angiography-derived FFR (angio-FFR) improved outcomes for PCI compared with a standard angiography-guided strategy.

Like FFR, angio-FFR is also performed in a binary manner to determine whether a vessel requires intervention and does not automatically indicate the haemodynamic improvement that would be expected post stenting. However, one advantage of angio-FFR is that virtual pullback could be generated during its calculation. Most importantly, though hyperemic blood flow was applied in angio-FFR calculation, it was predicted from resting flow with mathematical algorithm. As resting flow is more constant, consistent, and predictable across different stenoses, then resting pressure changes measured along the length of a vessel will be more predictable. Using this property, a physiological vessel map could be produced with angio-FFR by co-registration the pullback onto coronary angiogram, which not only highlight functional significant lesions and lesion locations, but also offer the possibility of prospective simple computerized virtual PCI to assess the potential hemodynamic impact before actual stent implantation.

In this regard, the investigators aim to calculate angio-FFR and to develop an angio-FFR pullback. And the investigators hypothesize that angio-FFR-derived pullback would be possible to produce a physiological map showing lesion severity and location, in addition, it could be used to perform virtual PCI and predict the physiological impact of stenting; the physiological map could be used to measure physiological lesion length and intensity.

ELIGIBILITY:
Inclusion Criteria:

* any patient meets eligible criteria who underwent PCI with DES followed by invasive physiologic assessment at the index procedure
* any patient who underwent PCI for lesions with pre-PCI FFR<=0.80
* available of both pre- and post-PCI FFR measurement
* available of both pre- and post-PCI angio-FFR calculation
* available of pre-PCI co-registration of angio-FFR with coronary angiogram

Exclusion Criteria:

* unavailable pre-PCI angio-FFR calculation and co-registration with coronary angiogram
* unavailable post-PCI angio-FFR calculation
* culprit vessel of acute coronary syndrome
* failed achieving TIMI 3 flow at the end of PCI
* left ventricular ejection fraction <30%
* graft vessel
* collateral feeder
* in-stent restenosis
* primary myocardial or valvular heart disease
* in patient whose life expectancy less than 2 years
* visible thrombus of target vessel segment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed obstructive coronary artery disease and evaluated by pre-PCI FFR measurement, then treated by DES with invasive physiologic evaluation at the index procedure.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Propotion of angio-FFR based physiological map successfully created | Immediate after angiography
  Propotion of successful angio-FFR based physiological map created by overlaying the angio-FFR based pullback onto coronary angiogram will be calculated
Correlation of predicted post-PCI angio-FFR by physiological map with angio-FFR after PCI | Immediate post-PCI
  Pearson Correlation analysis will be performed to assess the correlation of predicted post-PCI angio-FFR by physiological map with angio-FFR after PCI
Agreement of predicted post-PCI angio-FFR by physiological map with angio-FFR after PCI | Immediate post-PCI
  Bland-altman analysis will be performed to assess the agreement of predicted post-PCI angio-FFR by physiological map with angio-FFR after PCI

SECONDARY OUTCOMES:
Correlation of pre-PCI angio-FFR with pre-PCI FFR | Immediate after pre-PCI FFR measurement
  Pearson Correlation analysis will be performed to assess the correlation of pre-PCI angio-FFR with pre-PCI FFR
Agreement of pre-PCI angio-FFR with pre-PCI FFR | Immediate after pre-PCI FFR measurement
  Bland-altman analysis will be performed to assess the agreement of pre-PCI angio-FFR with pre-PCI FFR
Correlation of post-PCI angio-FFR with post-PCI FFR | Immediate post-PCI FFR measurement
  Pearson Correlation analysis will be performed to assess the correlation of post-PCI angio-FFR with post-PCI FFR
Agreement of post-PCI angio-FFR with post-PCI FFR | Immediate post-PCI FFR measurement
  Bland-altman analysis will be performed to assess the agreement of post-PCI angio-FFR with post-PCI FFR
Correlation of pre-PCI angio-FFR derived pullback pressure gradient (PPG) with post-PCI angio-FFR | Immediate post-PCI
  Pearson Correlation analysis will be performed to assess the correlation of pre-PCI angio-FFR derived pullback pressure gradient with post-PCI angio-FFR
Correlation of pre-PCI angio-FFR derived pullback pressure gradient with post-PCI FFR | Immediate post-PCI
  Pearson Correlation analysis will be performed to assess the correlation of pre-PCI angio-FFR derived pullback pressure gradient with post-PCI FFR
Target Vessel Failure | 2 years after index procedure
  a composite of cardiac death, clinical-driven target vessel-related myocardial infarction, and clinical-driven target vessel revascularization. The target vessel will be defined as the treated vessel with 2nd generation DES which was assessed by post-stenting fractional flow reserve.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dai N, Che W, Liu L, Zhang W, Yin G, Xu B, Xu Y, Duan S, Yu H, Li C, Yao K, Huang D, Ge J. Diagnostic Value of Angiography-Derived IMR for Coronary Microcirculation and Its Prognostic Implication After PCI. Front Cardiovasc Med. 2021 Oct 15;8:735743. doi: 10.3389/fcvm.2021.735743. eCollection 2021. PMID 34722667
- [Background] Shin D, Dai N, Lee SH, Choi KH, Lefieux A, Molony D, Hwang D, Kim HK, Jeon KH, Lee HJ, Jang HJ, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Doh JH, Shin ES, Nam CW, Koo BK, Gwon HC, Ge J, Lee JM. Physiological Distribution and Local Severity of Coronary Artery Disease and Outcomes After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1771-1785. doi: 10.1016/j.jcin.2021.06.013. PMID 34412795
- [Background] Dai N, Hwang D, Lee JM, Zhang J, Jeon KH, Paeng JC, Cheon GJ, Koo BK, Ge J. Feasibility of Quantitative Flow Ratio-Derived Pullback Pressure Gradient Index and Its Impact on Diagnostic Performance. JACC Cardiovasc Interv. 2021 Feb 8;14(3):353-355. doi: 10.1016/j.jcin.2020.10.036. No abstract available. PMID 33541549